CLINICAL TRIAL: NCT02620722
Title: A New Technique for Determining Limb Occlusion Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, James A. McEwen, Principal Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H14-02048
Record Dates: First submitted 2015-12-01; First posted 2015-12-03 (Estimated); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Tourniquet Safety and Effectiveness
Keywords: tourniquet; safety; personalized; surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LOP Measurement (Experimental): Measure the limb occlusion pressure in each patient using the new technique with the personalized tourniquet instrument and the gold-standard technique with the handheld Doppler ultrasound.
  Interventions: Device: Personalized Tourniquet Instrument; Device: Handheld Doppler ultrasound

INTERVENTIONS:
Device: Personalized Tourniquet Instrument — Measure the limb occlusion pressure in each patient using the new technique with the personalized tourniquet instrument.
Device: Handheld Doppler ultrasound — Measure the limb occlusion pressure in each patient using the gold-standard technique with the Doppler ultrasound.

SUMMARY:
This study evaluates a novel technique for measuring the minimum pressure necessary to achieve a bloodless surgical field, known as a patient's limb occlusion pressure (LOP). Patients will have tourniquets applied to their arms and legs and LOP will be measured using the new technique and a gold standard Doppler ultrasound technique.

DETAILED DESCRIPTION:
Optimal tourniquet safety depends on accurately determining the minimum pressure necessary to achieve a bloodless surgical field, known as a patient's limb occlusion pressure (LOP). However, LOP is not yet routinely measured in all patients due to limitations of current techniques. This study evaluates a novel technique for measuring the LOP through the tourniquet cuff that overcomes many limitations of current LOP measurement techniques.

The goal of the study is to determine if the LOP measured by the new technique is statistically or clinically different from the LOP measured by a gold standard Doppler ultrasound technique in adult and pediatric patients

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for a visit to one of four surgical clinics in Vancouver, Canada
* Agreed to participate in the study and provide informed consent

Exclusion Criteria:

* Unable to give informed consent on their own behalf or by a legal guardian
* Lack of parental agreement in the case of consent from a legally competent minor
* Standard contraindications to tourniquet use
* Vascular disease or circulation problems in the extremities
* History or indication of deep vein thrombosis

Ages: 3 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2014-09; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Limb Occlusion Pressure Measurement (mmHg) using the new technique and the gold-standard technique | at time of measurement

SECONDARY OUTCOMES:
Limb Occlusion Pressure Measurement (mmHg) using the new technique and the existing distal sensor-based technique | at time of measurement

CONTACTS AND LOCATIONS:
Overall Officials: James A McEwen, PhD, Principal Investigator — University of British Columbia
Locations (4):
- Canada (4):
  - Complex Joint Clinic, Vancouver General Hospital, Vancouver, British Columbia
  - Cambie Surgery Centre, Vancouver, British Columbia
  - Foot and Ankle Clinic, St. Paul's Hospital, Vancouver, British Columbia
  - BC Children's and Women's Hospital, Vancouver, British Columbia

REFERENCES:
- [Background] Noordin S, McEwen JA, Kragh JF Jr, Eisen A, Masri BA. Surgical tourniquets in orthopaedics. J Bone Joint Surg Am. 2009 Dec;91(12):2958-67. doi: 10.2106/JBJS.I.00634. PMID 19952261
- See also: Educational website about tourniquets — http://tourniquets.org/index.php